CLINICAL TRIAL: NCT06903156
Title: Prospective Multicentre, Randomized, Double-blind, Placebo-controlled, Parallel-group Comparative Trial of the Efficacy and Safety of Different Dosages in Sequential Therapy With Mexidol® in Patients With Primary Open-angle Glaucoma
Brief Title: Efficacy and Safety of Different Dosages of Mexidol® in Patients With Primary Open-angle Glaucoma (POAG)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pharmasoft (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MexidolPOAG2023; PHS-FOG-006-MEX-SOL-TAB (Other: Ministry of Health, Russian Federation)
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Primary Open-Angle Glaucoma (POAG)
Keywords: Glaucoma; Primary Open-Angle Glaucoma (POAG); Glaucomatous Optic Neuropathy (GON); Mitochondrial Dysfunction; Neuroprotection; Retiniprotection; Mexidol; Ethylmethylhydroxypyridine Succinate
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma; Mitochondrial Diseases | interventions — emoxypine succinate; ethylmethylhydroxypyridine succinate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mexidol High (Active Comparator): High dose of Mexidol (Mexidol IV 500 mg 1 time a day for 14 days, then Mexidol FORTE 250 orally 250 mg 1 tablet 3 times a day for 90 days) and standard therapy
  Interventions: Drug: Mexidol
- Mexidol Low (Active Comparator): Low dose of Mexidol (Mexidol IV 100 mg 1 time a day for 14 days, then Mexidol 125 mg 1 tablet 3 times a day for 90 days) and standard therapy
  Interventions: Drug: Mexidol
- Placebo (Placebo Comparator): Placebo and standard therapy according to a scheme similar to Mexidol groups
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Mexidol — Neuroretinoprotector
  Other Names: Ethylmethylhydroxypyridine Succinate
  Arms: Mexidol High; Mexidol Low
Other: Placebo — Placebo therapy
  Arms: Placebo

SUMMARY:
The present trial is planned to investigate and identify the best dosage of investigational drugs with respect to the treatment of open-angle glaucoma. Therefore, multiple dose regimens of the investigational drug versus placebo drug are anticipated.

DETAILED DESCRIPTION:
Glaucoma is a widespread group of diseases, which are united by disorders of the hydrodynamics of the eye with increased intraocular pressure (IOP), development of glaucoma optic neuropathy (GON) and corresponding irreversible changes in the optic nerve and visual fields.

The number of glaucoma patients worldwide ranges from 60.5 to 105 million, more than 1 million glaucoma patients have been identified in Russia, but it is assumed that the true number of patients is twice as high. According to epidemiological analysis, primary open-angle glaucoma (POAG) is the most common glaucoma worldwide, accounting for 75% to 90% of all primary glaucoma.

The active substance of Mexidol (ethylmethylhydroxypyridine succinate) has a multitarget effect on a number of links in the pathogenesis of POAG and is characterised by a high degree of safety, which corresponds to the concept of multimodal and modulating therapy of GON in POAG.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes aged 35 to 75 years inclusive.
* Diagnosis of primary open-angle glaucoma stage II or III in both eyes.
* Intraocular pressure (IOP) compliance with ""target level"": tonometric IOP <21 mmHg in stage II, <19 mmHg in stage III, in both eyes.
* The patient's willingness and ability to fulfil the requirements of the protocol throughout the trial.
* Patients who signed informed consent to participate in the trial.
* For women with preserved reproductive potential, a negative pregnancy test and agreement to use adequate contraceptive methods throughout the trial.
* For men, agreement to adhere to adequate contraceptive methods for the duration of trial participation.

Exclusion Criteria:

* Individual intolerance or hypersensitivity to any of the components of the investigational medicinal products according to anamnesis data.
* Administration of nootropic, vasoactive drugs, neuroprotectants, antioxidants, metabolic drugs for 30 days prior to randomisation.
* The need to use medications that are prohibited in this trial.
* Primary open-angle glaucoma stage I or IV in at least one eye.
* Closed-angle glaucoma of at least one eye.
* The only eye.
* Diagnosis of primary open-angle glaucoma stage II or III in one eye only.
* Visual acuity less than 0.1 (with correction) in at least one eye.
* Presence of an active infectious-inflammatory process in at least one eye.
* Low reliability of SAP results in at least one eye due to the patient's condition/disease: presence of 20% or more false positive and/or false negative errors, large amplitude and frequency of gaze direction deviations.
* The "mean deviation" (MD) score for static automatic perimetry (SAP) is -20 decibels or worse in at least one eye.
* Surgical and/or laser interventions on at least one eyeball within 3 months prior to inclusion in the trial.
* Significant opacities of the optical media in at least one eye, preventing assessment of the efficacy of therapy, including: severe scarring of the cornea, cataracts, consequences of uveitis.
* Retinal detachment in at least one eye.
* Thrombosis of a central retinal vein or artery in at least one eye.
* Myopia with a length of the anteroposterior axis of the eyeball greater than 26 mm in at least one eye.
* Diabetic retinopathy and other eye conditions that may affect the assessment of therapy efficacy.
* Presence of a history or finding of clinically significant pathology on screening, including but not limited to those listed below: unstable angina pectoris within 3 months before inclusion in the trial; myocardial infarction within 3 months prior to inclusion in the trial; acute heart failure; severe arrhythmia requiring treatment with class Ia, Ib, Ic or III antiarrhythmic drugs; decompensation of chronic heart failure (according to the New York Heart Association classification) within 3 months before inclusion in the trial; uncontrolled arterial hypertension with systolic blood pressure >180 mmHg and/or diastolic blood pressure >100 mmHg at screening; brain injury, stroke or transient ischaemic attack within 6 months prior to screening; occlusive blood vessel diseases; stenosing blood vessel diseases resulting in significant ischaemia of the relevant blood supply area; metabolic disorders, including severe renal insufficiency (creatinine clearance less than 30 ml/min); severe hepatic insufficiency (ALT or AST level is at least 2 times higher than the upper limit of normal values); malignant diseases of any localization with duration of remission less than 5 years according to anamnesis; II or III degree respiratory failure; community-acquired pneumonia within 6 months prior to inclusion in the trial; severe and/or uncontrolled endocrine and metabolic disorders requiring continuous medication; type 1 diabetes mellitus; type 2 diabetes mellitus, with a disease duration of 5 or more years; gastrointestinal disorders in the phase of relapse or exacerbation and requiring continuous medication.
* Positive serological reactions for infections at screening: Human immunodeficiency virus (antibodies to HIV-1/2); Hepatitis B (surface antigen); Hepatitis C (antibodies to hepatitis C virus antigens); Syphilis (antibodies to Treponema pallidum).
* Presence of other ophthalmological, neurological, otolaryngological or systemic diseases that may be the cause of optic nerve damage.
* The presence of any other pathology that, in the opinion of the investigator, is a contraindication to the patient's participation in the trial (i.e. may adversely affect the patient's condition if he or she participates in the trial), may interfere with the conduct of the trial procedures, or affect the ability to interpret the results of the trial. In case of doubt, the investigator should consult with the trial medical monitor.
* Signs of a first detected disease/pathology at screening.
* Positive rapid test for IgM antibodies to SARS-CoV-2 and/or positive SARS-CoV-2 RNA using nucleic acid amplification techniques
* Current or history (two years prior to screening) of alcoholism, drug abuse, drug dependence and/or substance abuse.
* Mental, physical and other reasons that make it impossible to adequately assess one's behaviour and correctly comply with the conditions of the trial protocol, including a history of mental illness.
* Lack of willingness to co-operate on the part of the patient.
* Pregnancy and breastfeeding period. A positive pregnancy test in women of childbearing potential.
* Patient participation in another clinical trial within the last 30 days.
* Patient refusal to continue participation in the trial.
* A decision by the Investigator or Sponsor to exclude a patient from the trial due to a significant protocol deviation/protocol violation.
* A serious adverse event (SAE) or an adverse event that does not meet the criteria for seriousness, for which, in the opinion of the Investigator, further participation in the trial may be detrimental to the health or well-being of the patient, or for which withdrawal of the investigational therapy is necessary.
* The need for procedures and/or adjunctive therapy not authorized by the protocol of this trial.
* Allergic reaction or individual intolerance to the investigational drugs, requiring their cancellation.
* Non-compliance with the therapy regime (patient's adherence to treatment with tablet form of the drug goes beyond 80%-120%, parenteral therapy - 100%), non-adherence (loss of contact with the patient with subsequent non-appearance at the visit, violation of visit dates, etc.).
* Need for modification of topical hypotensive therapy.
* Occurrence during the trial of conditions/diseases specified in the inclusion criteria.
* Any patient condition that, in the reasonable judgement of the investigator, requires the patient to be excluded from the trial.
* Erroneous inclusion.
* Positive pregnancy test in a trial participant.
* Positive rapid test for IgM antibodies to SARS-CoV-2 and/or positive SARS-CoV-2 RNA using nucleic acid amplification techniques.
* Erroneous unblinding of trial subject's treatment group.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-09-07 (Actual); Study Completion 2023-09-07 (Actual)

PRIMARY OUTCOMES:
Mean change in mean deviation (MD) in static automated perimetry (SAP) at the end of the course of therapy vs. baseline | Day 104

SECONDARY OUTCOMES:
Mean change in the mean deviation (MD) of static automated perimetry (SAP) 14, 45 and 75 days from the start of therapy vs. baseline | 14, 45 and 75 days
Mean change in pattern standard deviation (PSD) at static automated perimetry (SAP) 14, 45, 75 and 104 days from the start of therapy vs. baseline | 14, 45, 75 and 104 days
Change in the number of relative scotomas (first and second order), number of absolute scotomas after 14, 45, 75 and 104 days from the start of therapy vs. baseline | 14, 45, 75 and 104 days
Mean change in visual acuity according to visometry without correction after 14, 45, 75 and 104 days from the start of therapy vs. baseline | 14, 45, 75 and 104 days
Mean change in visual acuity according to visometry with correction after 14, 45, 75 and 104 days from the start of therapy vs. baseline | 14, 45, 75 and 104 days
Mean change in the value of the threshold of electrical sensitivity of the optic nerve after 14, 45, 75 and 104 days from the beginning of therapy vs. baseline | 14, 45, 75 and 104 days
Mean change in the value of the electrical lability of the optic nerve after 14, 45, 75 and 104 days from the start of therapy vs. baseline level | 14, 45, 75 and 104 days
Dynamics of changes severity according to optical coherence tomography data after 14, 45, 75 and 104 days from the beginning of therapy in comparison with the initial level | 14, 45, 75 and 104 days
Dynamics of the severity of changes according to Heidelberg retinal tomography data after 14, 45, 75 and 104 days from the start of therapy vs. baseline | 14, 45, 75 and 104 days

CONTACTS AND LOCATIONS:
Locations (7):
- Russia (7):
  - Kirov Regional State Budgetary Healthcare Institution "Kirov Clinical Ophthalmological Hospital", Kirov
  - Federal State Budgetary Educational Institution of Higher Education "Moscow State Medical and Dental Institute named after A.I. Evdokimov" of the Ministry of Health of the RF, Moscow
  - Federal State Autonomous Institution "Intersectoral Scientific and Technical Complex "Eye Microsurgery" named after Academician S.N. Fedorov" of the Ministry of Health of the RF, Moscow
  - Budgetary healthcare institution of the Omsk region "V.P. Vyhodtsev Clinical Ophthalmological Hospital", Omsk
  - Saint Petersburg State Budgetary Healthcare Institution "State Hospital No. 40 of the Kurortny District", Saint Petersburg
  - Private healthcare institution "Clinical hospital "RZhD-Medicine" of the city of Saratov", Saratov
  - State Budgetary Institution of Healthcare of the Yaroslavl Region "Clinical Hospital No. 2", Yaroslavl